CLINICAL TRIAL: NCT01024790
Title: Behavioral Activation Enhanced Exercise Intervention:Pre-Pilot
Brief Title: Exercise Study to Help Patients Who Have Type 2 Diabetes and Depression.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Kristin Schneider, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13269
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise group (Experimental)
  Interventions: Behavioral: Exercise group
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Exercise group — 24 week group exercise class supplemented with behavioral activation strategies
  Arms: Exercise group

SUMMARY:
The purpose of this study is to test an exercise treatment that includes behavioral strategies to improve blood sugar control in women with type 2 diabetes who are depressed and overweight.This research study may lead to a potentially useful treatment for diabetes management when depression is present.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes, depression, BMI <44,ages between 21-65, female

Exclusion Criteria:

* BMI >44, >100 min. of exercise per week, Type 1 diabetes, no diabetes,MI,Stroke, Catheterization, unstable angina in previous 6 months,pregnancy,glucocorticosteroid therapy in last 3 months,bipolar, psychotic disorder or post-traumatic disorder,moving out of area within next 6 weeks

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
This research study may lead to a potentially useful treatment for diabetes management when depression is present. | 6 weeks
HbA1c | 3-,6-, and 9-months
Depression | 3-, 6- and 9-months

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Schneider, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Background] Schneider KL, Pagoto SL, Handschin B, Panza E, Bakke S, Liu Q, Blendea M, Ockene IS, Ma Y. Design and methods for a pilot randomized clinical trial involving exercise and behavioral activation to treat comorbid type 2 diabetes and major depressive disorder. Ment Health Phys Act. 2011 Jun 1;4(1):13-21. doi: 10.1016/j.mhpa.2011.04.001. PMID 21765864